CLINICAL TRIAL: NCT02040168
Title: Evaluation of the Interest of a Nurse-implemented Sedation Protocol for the Reduction of the Duration of Mechanical Ventilation Complication Associated With Extended Sedation in Pediatric Intensive Care Unit.
Brief Title: Reduce Pediatric Sedation to Reduce Mechanical Ventilation Complication in ICU
Acronym: PEDIASED
Status: Completed | Type: Observational
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: PROG/10/53
Record Dates: First submitted 2013-11-26; First posted 2014-01-20 (Estimated); Last update posted 2021-09-16 (Actual); Status verified 2021-09

CONDITIONS: Mechanical Ventilation Complication
Keywords: Ventilation; PTSD; sedation
MeSH Terms: conditions — Respiratory Aspiration; Stress Disorders, Post-Traumatic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 28 days - 18 yo: Children requiring mechanical ventilation for at least 24h from 28 days to 18 yo
- 18 months - 18 yo: Post traumatic stress disorder evaluation in children requiring mechanical ventilation for at least 24h from 18 month to 18 Years old

SUMMARY:
Mechanical ventilation is a common procedure used in pediatric intensive care units (ICU). Its use requires almost always the establishment of a sedation. Sedation is a generic term for all procedures, pharmacological or not, ensuring physical and psychological comfort and the safety of patient admitted in intensive care units.

An inadequate sedation, insufficient or excessive, has common side effects, as increase of the duration of mechanical ventilation and of hospital-acquired infections (in particular, ventilator associated pneumonia), of hemodynamic disorders, of extubation failure or accidental extubation, of withdrawal syndrome, and of post-traumatic stress disorder (PTSD). All these complications increase mechanical ventilation time and ICU length of stay. Several studies in adult's population have shown that the implementation of a sedation algorithm allowed to decrease the incidence of these complications.

We hypothetized that the duration of mechanical ventilation would be reduced by a nurse-implemented sedative management protocol.

DETAILED DESCRIPTION:
1. During the first period (15 months), no protocol is used. This period consists to assess current analgesia-sedation procedure used in the pediatric intensive care unit (PICU), associated with the collection of medical and socio-demographical data about mechanical ventilation duration, sedation complications, PTSD development. The severity of pathology can be evaluated using PIM2 and POPC scores. The sedation deepness will be determined using COMFORT-B scale. Eight weeks after hospitalization, families will be phoned to assess children memories, anxious troubles, and PTSD symptoms for the patients of more than 18 months old.
2. During the transition period (6 months), nurses and physicians develop the protocol and undergo training in its use.

During the third period, a nurse-implemented sedation is used. The collected data are the same that the collected data during the first period

ELIGIBILITY:
Inclusion Criteria:

* Children aged 28 days to 18 years
* Admitted in pediatric intensive care unit
* Necessity of mechanical ventilation > 24 hours.

Exclusion Criteria:

* Sedation started in another intensive care unit > 24 hours

Ages: 28 Days to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The old children from 28 days to 18 years admitted in pediatric intensive care unit of Nantes University Hospital requiring mechanical ventilation for at least 24 hours can be included in this study.
Sampling Method: Non-Probability Sample
Enrollment: 106 (Actual)
Dates: Start 2010-10-01 (Actual); Primary Completion 2014-12-31 (Actual); Study Completion 2015-10-31 (Actual)

PRIMARY OUTCOMES:
Duration of the ventilation period | Hospitalization + 8 weeks
  30% decrease of the ventilation period

SECONDARY OUTCOMES:
evaluate the impact of sedation protocol on short-term consequences of prolonged sedation | Hospitalization + 8 weeks
  Hospitalization length reduction PTSD incidence reduction of 50% Weaning syndrom incidence decrease Sedation drugs total dose decrease Decrease of mechanical ventilation related infections Decrease of accidental or self extubation frequency Required amine total dose decrease Correlation between sedation level and PTSD frequency Analysis of PTSD risk factors

CONTACTS AND LOCATIONS:
Overall Officials: Liet Jean Michel, Principal Investigator — Nantes UH
Locations (1):
- Nantes University Hospital, Nantes, Loire-Atlantique, France